CLINICAL TRIAL: NCT07095868
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of EVM14 as Monotherapy and in Combination With Pembrolizumab in Patients With Selected Solid Tumors
Brief Title: Evaluate the Safety, Tolerability, and Preliminary Efficacy of EVM14 Alone and in Combination in Patients With Selected Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Everest Medicines (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Everest Medicines (China) Co.,Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EVM14C101
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Selected Types of Solid Tumor
Keywords: Solid Tumor; Cancer Vaccine
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase I Dose Escalation in Monotherapy Cohort (Experimental)
  Interventions: Biological: EVM14
- Phase I Dose Escalation in Combination Therapy Cohort (Experimental)
  Interventions: Biological: EVM14; Combination Product: Pembrolizumab
- Phase IIa Dose Level A for tumor type 1 (Experimental)
  Interventions: Biological: EVM14; Combination Product: Pembrolizumab
- Phase IIa Dose Level B for tumor type 1 (Experimental)
  Interventions: Biological: EVM14; Combination Product: Pembrolizumab
- Phase IIa Control arm for tumor type 1 (Active Comparator)
  Interventions: Combination Product: Pembrolizumab
- Phase IIa Combo therapy for tumor type 2 (Experimental)
  Interventions: Biological: EVM14; Combination Product: Pembrolizumab
- Phase IIa Control for tumor type 2 (Active Comparator): For patients with tumor type 2, pembrolizumab 200 mg alone will be administered intravenously (IV infusion) every 3 weeks (Q3W) if disease progression doesn't occur.
  Interventions: Combination Product: Pembrolizumab

INTERVENTIONS:
Biological: EVM14 — Cancer Vaccine
  Arms: Phase I Dose Escalation in Combination Therapy Cohort; Phase I Dose Escalation in Monotherapy Cohort; Phase IIa Combo therapy for tumor type 2; Phase IIa Dose Level A for tumor type 1; Phase IIa Dose Level B for tumor type 1
Combination Product: Pembrolizumab — Anti-PD1 antibody
  Arms: Phase I Dose Escalation in Combination Therapy Cohort; Phase IIa Combo therapy for tumor type 2; Phase IIa Control arm for tumor type 1; Phase IIa Control for tumor type 2; Phase IIa Dose Level A for tumor type 1; Phase IIa Dose Level B for tumor type 1

SUMMARY:
Brief Summary:

The purpose of this clinical trial is to evaluate the safety, tolerability, preliminary efficacy, and immunogenicity of EVM14 administered intramuscularly (IM) alone and in combination with pembrolizumab in patients with selected solid tumors.

DETAILED DESCRIPTION:
EVM14C101 study is a First in Human(FIH), open-label, multiregional, multicenter study conducted in 2 Phases: Phase I and Phase IIa. In Phase I, EVM14 will be administered intramuscularly(IM) as a monotherapy (Mono Cohort) and in combination with pembrolizumab (Combo Cohort) in patients with solid tumors to assess the safety and tolerability, immunogenicity, preliminary efficacy of EVM14 as monotherapy and in combination with pembrolizumab. Based on the safety and immunogenicity data of Phase I, dose of EVM14 will be selected for the Phase IIa. In Phase IIa, the safety and tolerability, preliminary efficacy, and immunogenicity of EVM14 in combination with pembrolizumab will be further assessed in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Selected types of solid tumor that are pathologically confirmed unresectable advanced, recurrent, or metastatic.
2. Patients with at least 1 evaluable lesion assessed by Investigators within 28 days prior to the first dose of study treatment as defined per RECIST v1.1.
3. Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1 at Screening.
4. Life expectancy ≥ 3 months.
5. Patients must have adequate organ function.
6. At screening, patients must agree to provide, if available, tumor tissue for biomarker analysis. When archival tumor tissue is not available, it is optional for the patient to undergo a fresh biopsy to collect tumor tissue if deemed medically safe by the Investigator.

Exclusion Criteria:

1. Has disease that is suitable for local treatment administered with curative intent.
2. Has a diagnosed and/or treated additional malignancy within 5 years prior to the first dose of study treatment except for: curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, and curatively resected in situ breast, cervical cancer, and prostate cancer.
3. Histologically/cytologically confirmed nasopharynx cancer. Has non-squamous histology NSCLC. If small cell elements are present, the patient is ineligible.
4. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
5. Has a diagnosis of immunodeficiency.
6. Use of systemic corticosteroid (> 10 mg/day prednisone or equivalent) or other immunosuppressive medication within 14 days before the first dose of study treatment.
7. Has active autoimmune disease that has required systemic treatment in past 2 years or history of autoimmune disease that has possibility of relapse or at risk of having these conditions.
8. Poorly controlled co-morbidity, including but not limited to poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg) and poorly controlled type 2 diabetes, or other serious conditions requiring systemic treatment. Active gastric or duodenal ulcer.
9. Cerebrovascular events (stroke, transient ischemic attack, etc.) within 6 months prior to the first dose of study treatment.
10. QTcF interval male > 450 msec; female > 470 msec Or serious cardiovascular disease within 6 months prior to the first dose of study treatment
11. The left ventricular ejection fraction (LVEF) < 50% during the screening period.
12. History of Stevens-Johnson syndrome or toxic epidermal necrolysis syndrome.
13. Patients known to be human immunodeficiency virus (HIV)-positive or have acquired immune deficiency syndrome (AIDS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Phase I and Phase IIa: Incidence and severity of adverse events | From the the start of the first dose of study treatment to 90 days after the last study treatment or new anti-cancer treatments started, whichever occurs earlier.
Phase I: Incidence of dose-limiting toxicities (DLT) | Mono cohort: 28-day period from the first EVM14 monotherapy dose. Combo cohort: Days 1 to 21: 21-day period from the first dose of EVM14 in combination with pembrolizumab.
Phase IIa tumor type 1: Progression-free survival (PFS) | From the baseline to disease progression confirmed by radiological examination, the start of a new anti-cancer treatment, withdrawal of informed consent, lost to follow-up, death, or end of study, whichever occurs first. (Up to 3 years)
  The time from date of randomization to the first documented disease progression per RECIST 1.1 evaluated by Investigators or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Phase I and Phase IIa: Objective response rate (ORR) | From the baseline to disease progression confirmed by radiological examination, the start of a new anti-cancer treatment, withdrawal of informed consent, lost to follow-up, death, or end of study, whichever occurs first. (Up to 3 years.)
  The percentage of patients meeting the criteria of best overall response as complete response (CR) or partial response (PR) evaluated by Investigators based on RECIST v1.1.
Phase I and Phase IIa: Disease control rate (DCR) | From the baseline to disease progression confirmed by radiological examination, the start of a new anti-cancer treatment, withdrawal of informed consent, lost to follow-up, death, or end of study, whichever occurs first. (Up to 3 years.)
  The percentage of patients meeting criteria of best overall response as stable disease (SD), PR, or CR evaluated by Investigators based on RECIST v1.1.
Phase I and Phase IIa: Duration of response (DOR) | From the baseline to disease progression confirmed by radiological examination, the start of a new anti-cancer treatment, withdrawal of informed consent, lost to follow-up, death, or end of study, whichever occurs first. (Up to 3 years.)
  The time between the date of earliest determination of CR or PR to the date of earliest documented progressive disease (PD), or to the date of death due to any cause, whichever occurs first.
Phase I and Phase IIa tumor type 2: Progression Free Survival (PFS) | From the baseline to disease progression confirmed by radiological examination, the start of a new anti-cancer treatment, withdrawal of informed consent, lost to follow-up, death, or end of study, whichever occurs first. (Up to 3 years.)
  The time from date of randomization or date of first dose to the first documented disease progression per RECIST 1.1 evaluated by Investigators or death due to any cause, whichever occurs first.
Phase IIa: Time to response (TTR) | From the baseline to disease progression confirmed by radiological examination, the start of a new anti-cancer treatment, withdrawal of informed consent, lost to follow-up, death, or end of study, whichever occurs first. (Up to 3 years.)
  The time between date of randomization/first dose and the date of first PR or CR.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, Fairfax, Virginia
- China (4):
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital With Nanjing Medical University, Nanjing, Jiangsu
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality